CLINICAL TRIAL: NCT07205172
Title: Gingival Phenotype and Dental Crowding in Pediatric Patients, a Pilot Study
Brief Title: Gingival Phenotype and Dental Crowding in Pediatric Patients
Acronym: BIOTIPO_PEDO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7704
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Crowding, Tooth; Gingival Diseases
MeSH Terms: conditions — Malocclusion; Gingival Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pediatric patients in the primary dentition stage: This group includes children who still have all their primary (baby) teeth, with no eruption of permanent teeth. Typically, this stage ranges from approximately 2 to 6 years of age.
  Interventions: Other: Orthodontic and periodontal analysis
- Pediatric patients in the early mixed dentition stage: This group includes children in the initial phase of tooth transition, where the first permanent molars and incisors have erupted while primary teeth are still present. This stage generally occurs between 6 and 8 years of age.
  Interventions: Other: Orthodontic and periodontal analysis
- Pediatric patients in the late mixed dentition stage: This group consists of children in the later phase of dental transition, when canines and premolars begin to replace primary teeth. It usually occurs between 9 and 12 years of age.
  Interventions: Other: Orthodontic and periodontal analysis
- Pediatric patients in the permanent dentition stage: This group includes adolescents who have completed the transition and have all or nearly all of their permanent teeth, excluding third molars (wisdom teeth). This stage typically begins around age 12 and up.
  Interventions: Other: Orthodontic and periodontal analysis

INTERVENTIONS:
Other: Orthodontic and periodontal analysis — Intraoral digital impression aimed at orthodontic analysis and periodontal evaluation using a dedicated periodontal probe, as part of the routine dental examination.

SUMMARY:
The diagnostic evaluation of the soft and hard tissues surrounding the tooth is one of the most crucial factors in clinical dental practice. It can influence treatment planning and decision-making in multidisciplinary dental care. Since different periodontal phenotypes respond differently to chemical, physical, and bacterial insults, or trauma during dental treatments, this aspect is considered essential in determining the outcome of therapy across many dental specialties.

Understanding the gingival phenotype can be of great importance in pediatric dentistry, as thick gingiva provides a solid and stable foundation for maintaining optimal oral hygiene and is one of the key elements in orthodontic treatment.

The bucco-lingual thickness of the gingiva, combined with the direction of tooth movement, is considered an important factor in soft tissue changes and in the development or progression of mucogingival defects. In cases of a thin phenotype, dehiscence and/or fenestrations may occur, predisposing the patient to gingival recession if the tooth is moved beyond the biological limits-i.e., outside the bony housing. The mandibular incisors have been identified as the teeth most susceptible to the development of labial recession.

Some malocclusions become evident as early as the early mixed dentition period. Intense changes in both soft and hard tissues occur during the growth and development of the stomatognathic system, as described in the literature, particularly during the mixed dentition phase. These changes can affect tooth position and the stability of periodontal tissues, making a proper evaluation of the gingival phenotype essential in pediatric patients.

Interceptive orthodontics plays a key role in the prevention and early management of malocclusions, helping to reduce the risk of developing mucogingival defects in adulthood. Early identification of a thin gingival phenotype allows for the implementation of preventive strategies, such as controlling tooth movement within biological limits and, if necessary, using gingival grafts before performing critical orthodontic movements.

Additionally, genetic, anatomical, and functional factors influence the gingival response to orthodontic forces. An accurate assessment of the gingival biotype, combined with personalized orthodontic planning, is essential to ensure effective treatment and long-term periodontal health.

Currently, there are no studies in the literature regarding the association between the severity of dental crowding and periodontal biotype in pediatric patients. Furthermore, the data available in the adult population are inconsistent: Kaya et al. demonstrated that, in adulthood, there is no correlation between the gingival phenotype and skeletal malocclusion. On the other hand, Kong et al. reported a correlation between a thin biotype in skeletal Class I and III, site-specific to the left mandibular central incisor, and also found a significant association between the thin phenotype and the normodivergent and hypodivergent groups.

To date, there is therefore no predictive model capable of identifying periodontal issues related to severe crowding.

The aim of this study is primarily to assess the periodontal phenotype in pediatric patients at different stages of dental transition and to investigate a possible association between a thin periodontal biotype and severe dental crowding in childhood.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients attending the Pediatric Dentistry and/or Orthodontics clinic (consultation and/or outpatient appointment).
* Parents and/or legal guardians have signed the informed consent for participation in the study.
* Age between 5 and 16 years.
* Clinical dentition criteria by group:

Group 1 (Primary Dentition): Presence in the mandibular arch of deciduous teeth from canine to canine. Group 2 (Early Mixed Dentition): Presence in the mandibular arch of at least two permanent mandibular incisors, fully erupted (incisal edge at occlusal level) or partially erupted (≥50% of the crown), with no clinical attachment loss, and healthy gingiva or mild gingivitis (Gingival Index, GI ≤ 1). Group 3 (Late Mixed Dentition): Presence in the mandibular arch of all four permanent mandibular incisors fully erupted (incisal edge at occlusal level), with no clinical attachment loss, and healthy gingiva or mild gingivitis (GI ≤

1). Group 4 (Permanent Dentition): Presence in the mandibular arch of all four permanent mandibular incisors fully erupted (incisal edge at occlusal level), with no clinical attachment loss, and healthy gingiva or mild gingivitis (GI ≤ 1).

Exclusion Criteria:

Patient-related:

* Parents and/or legal guardians have not signed the informed consent.
* Patients who are not sufficiently cooperative to allow a routine dental examination.
* Non-cooperative patients, including those with special needs.
* Children with systemic diseases or undergoing medication that affects gingival tissues.
* Patients who have already undergone orthodontic treatment or are currently undergoing orthodontic treatment.

Tooth-related:

* Presence of dental agenesis or dental anomalies.
* Dental sites with mucogingival problems.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric population of both sexes, aged between 5 and 16 years.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Gingival Phenotype in Pediatric Patients Across Dentition Stages | 24 months (18 months data collection, 12 months data processing and analysis)
  Assessment of gingival phenotype in pediatric patients categorized by dentition stage:
  Group 1: Primary dentition Group 2: Early mixed dentition Group 3: Late mixed dentition Group 4: Permanent dentition
  Gingival phenotype will be classified as thin or thick based on standardized clinical criteria.
  Measurement Tool:
  Transgingival probing using a periodontal probe (probe transparency method)
  Unit of Measure:
  Categorical variable: Thin vs. Thick gingival phenotype
  Gingival thickness measured in millimeters (mm), if quantitative assessment is used.

SECONDARY OUTCOMES:
Comparison of Crowding Indices and Periodontal Biotype | From ethics committee approval through 24 months (18 months data collection, 12 months data processing and analysis)
  Quantitative assessment of dental crowding in pediatric patients across the four dentition groups.
  Measurement Tool:
  Little's Irregularity Index and/or arch length-tooth size discrepancy measured on digital models
  Unit of Measure:
  Millimeters (mm) of crowding or Index score (numeric value, continuous)

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Gallenzi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS

IPD SHARING:
Plan to Share IPD: No